CLINICAL TRIAL: NCT02263378
Title: Ellagic Acid and Annona Muricata May Modulate the Immune Response to High Risk HPV Infection. A Randomized, Controlled Trial.
Brief Title: A New Supplement for the Immune Response to HPV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, associate professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OASIT-K
Record Dates: First submitted 2014-07-17; First posted 2014-10-13 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: HPV Infection
Keywords: HPV, L-SIL
MeSH Terms: conditions — Papillomavirus Infections | interventions — Ellagic Acid

ARMS (2):
- supplement (Experimental)
  Interventions: Drug: ellagic acid + annona muricata
- not intervention (Placebo Comparator)
  Interventions: Drug: ellagic acid + annona muricata

INTERVENTIONS:
Drug: ellagic acid + annona muricata — pills

SUMMARY:
The purpose of this study is to evaluate whether a supplement in which ellagic acid plus annona muricata are combined, may modulate the immune response to high risk HPV infection. Sixty women will be enrolled in a randomized, controlled study, having a histological diagnosis of L-SIL correlated with high rish HPV types infection. Main outcome measure is the activation of onco suppressor protein by the supplement and secondary outcome is the clearance of HPV infection in the treated group.

ELIGIBILITY:
Inclusion Criteria:

* women with high risk HPV infection
* histological diagnosis of L-SIL

Exclusion Criteria:

* women with no high risk HPV infection
* women without histological diagnosis of L-SIL

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
variation of onco suppressor protein expression from basal values. The expression variations are represented by the different percentage of positive cells | 6 months

SECONDARY OUTCOMES:
clearance of the HPV infection | 6 months